CLINICAL TRIAL: NCT05880277
Title: Diagnostic Point of Care Ultrasound of Patellar Tendon in Female Collegiate Athletes
Brief Title: Diagnostic POCUS of Patellar Tendinopathy in Female Athletes
Acronym: POCUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Morgan Bagley, Assistant Professor, Youngstown State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YoungstownSU
Record Dates: First submitted 2023-05-03; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Patellofemoral Disorder
Keywords: POCUS

STUDY DESIGN:
Intervention Model Description: female collegiate jumping athletes
Masking Description: Team physician will exam images but will be blinded from participant. Will only see participant number.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Jumping (Experimental): Female jumping collegiate athletes
  Interventions: Diagnostic Test: POCUS

INTERVENTIONS:
Diagnostic Test: POCUS — Point of Care Ultrasound

SUMMARY:
Purpose: The purpose of this study is to determine the clinical effectiveness of point-of-care diagnostic ultrasound in the assessment of patellar tendon pathologies

DETAILED DESCRIPTION:
Participants will receive information about the study and informed consent will be provided. Participants will voluntarily agree to be a participant in the study. Participants will sign the informed consent, and complete the POCUS demographic information sheet, if they qualify then they will have both of their patellar tendons examined through the use of the Butterfly IQ diagnostic ultrasound. Following the examination, they will complete the Knee Injury and Osteoarthritis Outcome Score (KOOS) and the Knee Injury and Osteoarthritis Outcome Patellofemoral subscale (KOOS-PF) and then complete the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 yr. old female student-athletes who participate in jump-centric activities

Exclusion Criteria:

* anyone who does not fit the inclusion criteria (18-25 yr old female student-athletes who participate in jump-centric activities

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Changes of patellar tendons in jumping athletes | 2 years
  % of participants with hyperechoic or hypoechoic changes
KOOS | 2 years
  % of participants with hyperechoic or hypoechoic changes in relation to the Knee Injury and Osteoarthritis Scores

CONTACTS AND LOCATIONS:
Overall Officials: Morgan C Bagley, PhD, Principal Investigator — Faculty
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No